CLINICAL TRIAL: NCT01145287
Title: Impact of the Diagnosis of Celiac Disease
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Finnish Celiac Society (Unknown)
Responsible Party: Principal Investigator, Kalle Kurppa, M.D, pH.D, Pediatrician, Tampere University Hospital
Other Study IDs: Burden-1
Record Dates: First submitted 2010-06-07; First posted 2010-06-16 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Gluten-free diet; Screen-detected; Asymptomatic; Quality of life; Self-perceived health; Healthcare resource utilization
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this study is to assess the impact of the diagnosis of celiac disease on general health, healthcare resource utilization, quality of life and lifestyle. We hypothesize that diagnosis and subsequent dietary treatment may have positive impact on these variables.

DETAILED DESCRIPTION:
All new members with biopsy-proven celiac disease joining the Finnish Celiac Society will be categorized in three groups according to symptoms and signs leading to the diagnosis as classical symptoms, extraintestinal symptoms and screen-detected, the latest being further divided to those presenting with symptoms and those who are totally asymptomatic. Several parameters assessing general health and well-being, quality of life and healthcare resource utilization are evaluated at baseline and after one and five years on trial. Quality of life is compared to that of non-celiac controls.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis within one year
* biopsy-proven diagnosis

Exclusion Criteria:

* Celiac disease diagnosis previously than within one year
* No biopsy-proven diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All new members with biopsy-proven celiac disease joining the Finnish Celiac Society.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2007-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Psychological General Well-Being (PGWB) Index | 5 years
  Health-related quality of life and self-perceived health are evaluated at diagnosis and after five years on dietary treatment by using structured questionnaire

SECONDARY OUTCOMES:
healthcare resource utilization | 5 years
  Healthcare resuorce utilization measured as inpatient and outpatient visits and consumption of other medical services in addition to consumption of pharmaceutical agents
Gastrointestinal Symptoms Rating Scale (GSRS) | 5 years
  clinical symptoms are evaluated at diagnosis and after five years on dietary treatment by using structured questionnaire
dietary compliance | 5 years
  self-assessed compliance to the dietary treatment
weight | 5 years
  effect of the dietary treatment in the weight of celiac disease patients
height | 5 years
  effect of the dietary treatment in the height of children with celiac disease
The Short Form (SF-36) Health Survey | 5 years
  Health-related quality of life and self-perceived health are evaluated at diagnosis and after five years on dietary treatment by using structured questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Research Centre, University of Tampere, Tampere University Hospital, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Derived] Ukkola A, Kurppa K, Collin P, Huhtala H, Forma L, Kekkonen L, Maki M, Kaukinen K. Use of health care services and pharmaceutical agents in coeliac disease: a prospective nationwide study. BMC Gastroenterol. 2012 Sep 27;12:136. doi: 10.1186/1471-230X-12-136. PMID 23016889
- [Derived] Kinos S, Kurppa K, Ukkola A, Collin P, Lahdeaho ML, Huhtala H, Kekkonen L, Maki M, Kaukinen K. Burden of illness in screen-detected children with celiac disease and their families. J Pediatr Gastroenterol Nutr. 2012 Oct;55(4):412-6. doi: 10.1097/MPG.0b013e31825f18ff. PMID 22614110
- [Derived] Ukkola A, Maki M, Kurppa K, Collin P, Huhtala H, Kekkonen L, Kaukinen K. Changes in body mass index on a gluten-free diet in coeliac disease: a nationwide study. Eur J Intern Med. 2012 Jun;23(4):384-8. doi: 10.1016/j.ejim.2011.12.012. Epub 2012 Jan 28. PMID 22560391
- [Derived] Ukkola A, Maki M, Kurppa K, Collin P, Huhtala H, Kekkonen L, Kaukinen K. Patients' experiences and perceptions of living with coeliac disease - implications for optimizing care. J Gastrointestin Liver Dis. 2012 Mar;21(1):17-22. PMID 22457855